CLINICAL TRIAL: NCT02659267
Title: Evaluation of a Strategy Designed to Promote Physical and Healthy Eating Between Users of the Health Academy Program in Belo Horizonte, Minas Gerais - "VAMOS BEAGÁ"
Brief Title: Evaluation of a Strategy Designed to Promote Physical and Healthy Eating
Acronym: VAMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Simone Teresinha Meurer, PHD student, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VAMOS Beagá
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Health Promotion; Physical Activity; Eating habits; Health System; Users from Health Academy Program
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventions Group= (Experimental): Group of change behavior including physical activity and healthy eating habits promotion.
  Interventions: Behavioral: Interventions Group
- Control Group= (No Intervention): Group that will not receive the VAMOS program as intervention, only participate in the Health Academy Program Activities.

INTERVENTIONS:
Behavioral: Interventions Group — VAMOS is a lifestyle promotion strategy, designed to promote physical activity and healthy eating habits. The intervention is composed by a weekly meeting, 12-week, in group, lasting about 60 min. In each weekly meeting, were discussed guidelines and strategies for physical activities practices in different domains and for adoption of a healthy diet. All aspects and strategies included in the VAMOS strategy are based in behavior changes theories. The participants of this group received educational material and, in the middle of the program, they received a pedometer to aid in motivation and in the self-monitoring physical activity.
  Other Names: VAMOS
  Arms: Interventions Group=

SUMMARY:
The study aims to verify if the VAMOS strategy contributes to an increase in physical activity and healthy eating habits among users of the Health Academy Program from Belo Horizonte, Minas Gerais.

DETAILED DESCRIPTION:
The Health Academy Program (AP) is a important policy to promote physical activity in Brazil. There are areas with infrastructure, equipment, and human resources to stimulate and guide people doing physical activity in community settings at no cost. The study aims to verify if the VAMOS strategy contributes to an increase in physical activity and healthy eating habits among users of the Health Academy Program (AP) at Belo Horizonte, Minas Gerais - "VAMOS BEAGÁ". Two AP poles, both belonging the same regional administration of the municipality and with the same health vulnerability index were selected. To define the location of the intervention VAMOS was carried draw between the selected centers, and all potentially eligible users invited to participate. Users of the Intervention Group (IG) took part in the daily activities offered by AP and, additionally, for 12 weeks, they attended the educational strategy called VAMOS. The Control Group does only the regular activities of AP. The VAMOS has been evaluated by the dimensions of Reach, Effectiveness, Adoption (at the individual level), Implementation and Maintenance (at individual and organizational level) of the RE-AIM model (Reach, Efficacy / Effectiveness, Adoption, Implementation, Maintenance). The reach is evaluated by the rate of participation and representation among participants and those invited to join the VAMOS. The effectiveness has been evaluated from anthropometric measurements, eating habits, physical activity level, stages of change, self-efficacy, social support and quality of life before and after 12 weeks of intervention. To assess the adoption was investigated the interest of Physical Activity professional from AP in mediating this strategy in future. The implementation was evaluated by identifying the extent to which the VAMOS was conducted as planned. The maintenance, at individual level, will be estimated from revaluations of all outcomes, as measured before and after the intervention, sixs months after the conclusion of the intervention. At organizational level, the maintenance will be accessed with semi-structured interviews conducted with the coordinators and managers of AP assessed feasibility of continuing of VAMOS strategy in AP. For the analysis of qualitative data will be conducted content analysis. And to the quantitative data, we carried out descriptive statistics, paired tests chi-square or Fisher's exact and two-way ANOVA for repeated measures or Wilcoxon signed rank test. Intent-to-treat analyzes were used. The significance level was 5% and the statistical program used was the Statistical Package for Social Sciences (SPSS) for Windows.

The overall goal of this study is to evaluate a strategy to promote physical activity and healthy eating, called VAMOS, among users of the Health Academy Program in Belo Horizonte, Minas Gerais.

Specific objectives:

1. Evaluate the effectiveness of VAMOS strategy on the level of habitual physical activity, dietary profile and nutritional status of the participants;
2. To identify associations between psychosocial mediators of behavior - self-efficacy and social support - and changes in physical activity and dietary profile of the participants;
3. Analyze the VAMOS strategy regarding the effectiveness, adoption (at individual level), reach, implementation and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Must be user of de Health Academy Program selected for the survey;
* Must have 20 years or older;

Exclusion Criteria:

* Not agree to participated with study;
* Not agree to sign the written informed consent;

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change in physical activity | baseline, 12 weeks, 36 weeks
  Habitual physical activity has been assessed by GT3X or GT3X+ accelerometer (Actigraph - USA) and analysed with Actilife 6.10 software. Each participant was instructed to use the accelerometer on his/her waist for seven consecutive days, removing it only when sleeping, bathing or performing water activities. Attached to an elastic belt, the device had to stay at the right side of the hip. Data are recorded in a 30 Hz sample frequency and analyzed using 60-s epochs. Periods with consecutive values of zero (with 2-min of spike tolerance) for 60 min or longer are interpreted as "accelerometer not worn" and therefore excluded. Physical activity data are included only if the participant got a minimum of 10 hours/day of recording for at least four days, including at least one weekend day
change in frequency of consumption of fresh and minimally processed food | baseline, 12 weeks, 36 weeks
  The frequency of consumption of raw and cooked vegetables, fruits, milk, pulses, meat, fish and tubers / roots has been monitored. The following scores are assigned by means of questionnaire: daily consumption = 4 points; weekly consumption = 3 points, monthly consumption = 2 points; rare consumption= 1 point; null consumption = 0 point. Higher the resulting score, healthier the consumption.
change in Body mass index | baseline, 12 weeks, 36 weeks
  Body mass has been measured while participants wear light clothes and no shoes, using an automatic scale (Welmy - Brazil) to the nearest 0.1 kg. Height has been measured using a stadiometer connected to scale to the nearest 0.5 cm. Body mass index has been calculated as the ratio between body mass in kilograms and the square of height in meters.
change in waist circumference | baseline, 12 weeks, 36 weeks
  Waist circumference is measured at the lesser curvature identified between the last rib and the iliac crest.
change in hip circumference | baseline, 12 weeks, 36 weeks
  Hip circumference is measured in the area of larger diameter of the hip, without compressing the skin.
change in consumption of Ultra-Processed food | baseline, 12 weeks, 36 weeks
  The frequency of consumption of sausages, sandwich cookies, candy, snacks / fatty snacks, soda, juice powder and industrialized seasoning has been monitored. The following scores are assigned by means of questionnaire: daily consumption = 0 points; weekly consumption= 1 point; monthly consumption = 2 points, rare consumption = 3 points; null consumption = 4 points. Higher the resulting score, healthier the consumption.

SECONDARY OUTCOMES:
change in stages of self-changes for physical activity | baseline, 12 weeks, 36 weeks
  The stages of self-changes for physical activity are assessed by questionnaires that sort subjects in one of five stages: pre-contemplation, contemplation, preparation, action and maintenance.
change in stages of self-changes for healthy eating habits | baseline, 12 weeks, 36 weeks
  The stages of self-changes for healthy eating habits are assessed by questionnaires that classified subjects in one of five stages: pre-contemplation, contemplation, preparation, action and maintenance.
change in self-efficacy | baseline, 12 weeks
  The self-efficacy are evaluated by scale "Self-Efficacy to Regulate Eating Habits and Self-Efficacy to Regulate Exercise" proposed by Bandura (2006) and validated for Brazilian adults by Boff (2012).
change in social support | baseline, 12 weeks
  The social support for physical activities has been evaluated by a scale proposed by Reis et al. (2011).
change in quality of life | baseline, 12 weeks, 36 weeks
  The quality of life is assessed by two general questions from Whoqol BREF.

CONTACTS AND LOCATIONS:
Overall Officials: Tânia Rosane B Benedetti, Doctor, Study Director — Federal University of Santa Catarina; Aline Cristine S Lopes, Doctor, Study Director — Federal University of Minas Gerais; Simone T Meurer, PHD Student, Principal Investigator — Federal University of Santa Catarina
Locations (1):
- Simone Teresinha Meurer, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BOFF, R. de M. Evidências Psicométricas das Escalas de Auto-eficácia para regular hábito alimentar e Auto-eficácia para regular exercício físico. Dissertação (mestrado). Pontífica Universidade Católica do Rio Grande do Sul, Porto Alegre, 2012.
- [Background] Reis MS, Reis RS, Hallal PC. Validity and reliability of a physical activity social support assessment scale. Rev Saude Publica. 2011 Apr;45(2):294-301. doi: 10.1590/s0034-89102011000200008. English, Portuguese. PMID 21412569
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154